CLINICAL TRIAL: NCT02515591
Title: Validating the Use of Disposable Flexible Intubation Bronchoscopes for Research Bronchoalveolar Lavage
Brief Title: Validating the Use of Disposable Bronchoscopes for Research Bronchoalveolar Lavage
Acronym: BALval
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 15/NW/0019
Record Dates: First submitted 2015-07-21; First posted 2015-08-05 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Healthy volunteer; Respiratory; Bronchoalveolar lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage cells Bronchoalveolar lavage supernatent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bronchoalveolar Lavage validation study — Bronchoalveolar lavage involved the washing out of the right middle lobe of the lung of a healthy volunteer with 200mls of warmed normal saline with or without sedation.

SUMMARY:
Validation study to use the disposable bronchoscopes in healthy volunteer research bronchoscopies to ensure adequate sample and cell yield.

DETAILED DESCRIPTION:
Research bronchoscopies are traditionally performed using conventional flexible fibreoptic bronchoscopes. The technique for obtaining bronchoalveolar lavage fluid (BAL) from healthy volunteers for research purposes has been developed by our group since 1999 and has been performed in > 1,000 subjects in the UK and Malawi including healthy volunteers.

Fibreoptic bronchoscopy with BAL using manual hand held suction enables the removal of non-adherent cells and lung lining fluid from the mucosal surface. In research environments, BAL allows sampling of innate (lung macrophage), cellular (B- and T- cells), and humoral (immunoglobulin) responses within the lung. Further applications include determining protein and drug levels, with the latter being a key parameter in early phase 'lung tissue active' drug development.

The BAL technique uses gentle hand-held suction of instilled fluid; this is designed to maximize BAL volume returned, and to apply minimum shear force on ciliated epithelia in order to preserve the structure and function of cells within the BAL fluid. This technique is also intended to preserve viability to facilitate the growth of cells in ex vivo culture. The research technique therefore uses a larger volume of warmed normal saline instillate (typically in the order of 200 ml) and employs manual suction to reduce cell damage.

At the Royal Liverpool Hospital (RLBUHT) ≥120 healthy volunteer BALs have been performed. Available data suggest that from 200 ml of instillate the following volume yields are retrieved: mean 100-120 ml, median 120 - 125 ml with ~ 19% of BALs returning <100 ml yield. The preferable BAL volume yield is >100 ml, a yield of >150 ml is considered excellent; yields >170 ml have not been recorded. There is no linear relationship between the cell yield and volume yield. Yields of <100 ml are in our experience, more likely to lead to side effects such as cough, chest pain and fever. Subjects with yields of <100 ml are advised to be recovered in the left lateral position to aid postural drainage of remaining instillate. There have been no serious adverse events (SAEs) reported; and notably there have been no post procedure hospitalisations or antibiotics required for suspected pneumonia.

Single-use flexible intubation bronchoscopes are used throughout United Kingdom (UK) National Health Service (NHS) trusts. They are predominantly used within the intensive care and anaesthetic (theatre) setting for both emergency and elective airway intubation. The flexible fibreoptic bronchoscope with sterile single-use disposable-sheath endoscope system has the potential to be more cost-effective and reduce the risk, however negligible, of cross-infection during the sterilisation procedure. Eliminating the need for high-level disinfection processing between procedures reduces maintenance costs (equipment and staff), and scope downtime and provides the flexibility more suited for research in healthy volunteers.

The content of this study proposal has been peer reviewed by two senior research associates based in Malawi and the UK who have deemed the scientific review criteria to be sound.

Currently many new drug and therapeutics discovery and development projects are blighted by the absence of robust predictive pre-clinical models. For example, promising anti-tuberculosis (TB) drugs and drug combinations have been clinically trialled based on current in vitro and in vivo models, only to find that they lack clinical efficacy; and conversely effective anti-TB drugs such as linezolid had poor or modest efficacy in testing usingin vitro and in vivo models. To mitigate these issues we have therefore developed dynamic pharmacodynamic in vitro models based on high content imaging that are able to measure macrophage intracellular tubercular growth and killing rates. Pharmacodynamic (PD) and Pharmacokinetics (PK) modelling of these models more closely resemble clinical measurements for known first line anti-TB; therefore we now wish to further develop this platform into a more physiological model by using alveolar macrophages (AMs) obtained from human subjects.

The purpose of using human AMs will be to compare the drug effects of known and new anti-TB compounds in human AMs to other in vitro models. This work will enable us to obtain better, more clinically relevant parameters to predict the outcome of drug dynamics. By using the AMswe can assess how reliable our current model systems are, and assess considerations of drug action in clinically relevant tissue samples. These cells can then be manipulated ex vivo to desired clinical scenarios e.g. dual TB and HIV-infections monitoring TB responses over time to a range of novel drugs and novel drug combinations. The outputs of these studies will be used directly to inform new clinical trials on drug regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to provide written consent before any study procedures are performed and can understand and comply with the requirements of the study.
2. Males and non-pregnant females, between 18 and 55 years of age, inclusive.
3. Body mass index (BMI) 18.0 to 30.0 kg/m2, inclusive.
4. Fluent in English, ability to understand the procedures and convey any adverse events effectively to the research team.

Exclusion Criteria:

1. Subjects with hepatic, pulmonary, metabolic, neurologic, cardiovascular, gastrointestinal, haematological, or psychiatric system, or any significant condition that may preclude nasal or oral intubation with a bronchoscope ,in the opinion of the investigator.
2. Subjects with any report of acute illness or febrile event that has not resolved 72 hours before bronchoscopy.
3. Subjects with any use of, or intent to use, medications, including prescription, over the counter, herbal preparations, or vitamin/mineral supplementation, for 3 days before the bronchoscopy with the exception of contraception medication.
4. Subjects who have had previous adverse reactions to benzodiazepines or anaesthetic agents (lidocaine) including reversal agents such as flumazenil.
5. Subjects who have participated (taken investigative drug and/or device) in another clinical trial within 30 days or within drug's 5 half-lives, whichever is longer, before the study procedure.
6. Subjects with any elevation of liver test results above 2 times the upper limit of normal; isolated elevation of bilirubin levels without elevation of direct bilirubin level is acceptable.
7. Subjects with a haemoglobin level <12.0 g/dL and prothrombin time < 13 seconds.
8. Subjects with very poor venous access.
9. Subjects who have used cigarettes (including vapour / e-cigarettes), cigars, and nicotine-containing products within 3 months before bronchoscopy and have a smoking history of >10 pack years.
10. Subjects who have not abstained from alcoholic beverages or alcohol-containing products for at least 72 hours before bronchoscopy.
11. Female subjects with a positive urine pregnancy test at screen and/or prior to bronchoscopy.
12. Subjects who are employees of the study unit or their close family members, students who are working in the study unit, or close family members of the investigator or sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers, male and Non pregnant female, aged between 18-55 years old.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Volume Retrieved | Immediately post-bronchoscopy. Assessed at LSTM upon receipt. Up to 2 hours post bronchoscopy
  Yield-ml
Cell Yield and Viability | Immediate retrieval. Assessed at LSTM upon receipt. Up to 4hours post bronchoscopy
  Cell yield and viability (Total cell count and differential cell count of alveolar macrophages [AMs] and lymphocytes)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool Hospital Clinical Research Facility, Liverpool, United Kingdom

REFERENCES:
- [Derived] Zaidi SR, Collins AM, Mitsi E, Reine J, Davies K, Wright AD, Owugha J, Fitzgerald R, Ganguli A, Gordon SB, Ferreira DM, Rylance J. Single use and conventional bronchoscopes for Broncho alveolar lavage (BAL) in research: a comparative study (NCT 02515591). BMC Pulm Med. 2017 May 5;17(1):83. doi: 10.1186/s12890-017-0421-7. PMID 28476111